CLINICAL TRIAL: NCT05146089
Title: Reflex Responses to Intermittent Hypoxia in Humans: Mechanisms and Consequences
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007973; K99HL130339 (NIH); R00HL130339 (NIH)
Record Dates: First submitted 2021-11-02; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Sleep Apnea; Healthy; Vasoconstriction; Vasodilation
MeSH Terms: conditions — Sleep Apnea Syndromes; Aneurysm | interventions — Bosentan

STUDY DESIGN:
Intervention Model Description: Subjects will be asked to complete 1 1-hour screening visit, 1 overnight at-home monitoring, and 1 (women) or 2 (men) 5-hour study visits. Subjects will not be blinded to study condition and all subjects will serve as their own controls. All study visits will be separated by a minimum of 1 week and will occur at the same time of day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hypoxia Exposure (Experimental): Men and women will be exposed to acute intermittent hypoxic episodes.
  Interventions: Other: Hypoxic exposure; Other: modified Oxford test; Drug: Oral Bosentan 62.5 mg; Other: Hypoxic ventilatory response test

INTERVENTIONS:
Other: Hypoxic exposure — 30 minutes of intermittent hypoxia achieved using breaths of low oxygen air (5% oxygen) followed by room air through a mask.
Other: modified Oxford test — An intravenous bolus of sodium nitroprusside (100 μg) will be given to decrease blood pressure, followed 1 minute later by a bolus of phenylephrine (150 μg) to increase blood pressure, occurring before and after intermittent hypoxia exposure.
Drug: Oral Bosentan 62.5 mg — Prior to completion of visit 2, male subjects will consume 62.5 mg twice daily for 3 days as well as the morning of the study visit (7 pills) at home and experimental sessions will be performed 3 hours after oral intake of the final dose.
Other: Hypoxic ventilatory response test — Hypoxia will be achieved using breaths of low oxygen air (5% oxygen) followed by room air through a mask. This will be repeated 4-5 times per test, occurring before and after intermittent hypoxia exposure.

SUMMARY:
The overall goal of this project is to better understand the effect of intermittent hypoxia (IH) on sympathetic neuronal discharge patterns in humans, as well as mechanisms that mediate persistent sympathoexcitation with IH.

DETAILED DESCRIPTION:
Sleep apnea is the most common form of sleep disordered breathing and patients with sleep apnea exhibit persistent activation of the sympathetic nervous system. Sympathoexcitation is also the final common pathway for a host of complications in conditions like obesity, hypertension, sleep apnea, and heart failure and plays a significant role in predicting negative clinical outcomes and deteriorating cardiovascular health. However, the mechanisms of sympathoexcitation with sleep apnea are poorly understood and thus make effective therapeutic approaches difficult to develop.

Intermittent hypoxia (IH) has been implicated in animal models as the primary stimulus for evoking increases in sympathetic activity with recurrent apneas. Thus, the overall goal of this application is to better understand the effect of IH on sympathetic discharge patterns in humans as well as the mechanisms mediating persistent sympathoexcitation with IH. By better understanding the effect of IH on sympathoexcitation, targeted therapeutic approaches might be devised to mitigate the effects of sympathetic over-activity on the cardiovascular system in conditions such as sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult men and women;
* 18-45 years of age;
* BMI <30 kg/m2;
* non-pregnant/non-breastfeeding;
* non-smokers.

Exclusion Criteria:

Subjects will be excluded if they are:

* taking any medications known to affect the cardiovascular or autonomic nervous system (e.g. alpha-blockers, beta-blockers, etc);
* Apnea Hypopnea Index >10 events/hr

Self-reported history of:

* hepatic, renal, pulmonary, cardiovascular, or neurological disease;
* stroke or neurovascular disease;
* bleeding/clotting disorders;
* sleep apnea or other sleep disorders;
* diabetes;
* smoking;
* history of alcoholism or substance abuse;
* hypertension.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity (MSNA) | Change from baseline after hypoxia exposure
  MSNA burst incidence (bursts/100 heart beats)

SECONDARY OUTCOMES:
Arterial blood pressure | Change from baseline after hypoxia exposure
  Systolic blood pressure, Diastolic blood pressure, Mean blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline K Limberg, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - University of Missouri-Columbia, Columbia, Missouri
  - Mayo Clinic, Rochester, Missouri

IPD SHARING:
Plan to Share IPD: Undecided